CLINICAL TRIAL: NCT07265271
Title: A Cell-Free tsRNA-Based Liquid Biopsy Signature for Early Detection of Hepatocellular Carcinoma
Brief Title: A Cell-free tsRNA Signature for Early Detection of Hepatocellular Carcinoma
Acronym: CENTINEL
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/CENTINEL
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; Liver cancer; tsRNA; Liquid Biopsy; Early Detection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HCC (Discovery, Small RNA-seq): Serum and plasma samples from patients with histologically confirmed HCC will be analyzed using small RNA sequencing to identify circulating tsRNAs specifically upregulated in HCC. These tsRNAs will serve as candidates for downstream validation.
  Interventions: Diagnostic Test: Small RNA sequence
- Non-disease Control (Discovery, Small RNA-seq): Serum and plasma samples from individuals without malignant will be analyzed in parallel by small RNA sequencing to identify tsRNAs differentially expressed between HCC and non-disease controls.
  Interventions: Diagnostic Test: Small RNA sequence
- HCC (Training, rt-qPCR): Serum and plasma samples from patients with histologically confirmed HCC will be analyzed using rt-qPCR to test circulating tsRNAs specifically upregulated in HCC.
  Interventions: Diagnostic Test: Rt-qPCR
- NDC (Training, rt-qPCR): Individuals without malignant whose serum/plasma samples will serve as controls to establish baseline tsRNA expression and diagnostic thresholds.
  Interventions: Diagnostic Test: Rt-qPCR
- HCC (Testing, rt-qPCR): Independent HCC cohort used for external validation of the panel to confirm diagnostic performance and reproducibility.
  Interventions: Diagnostic Test: Rt-qPCR
- NDC (Testing, rt-qPCR): Individuals without malignant whose serum/plasma samples will be used for validation of specificity and model robustness.
  Interventions: Diagnostic Test: Rt-qPCR

INTERVENTIONS:
Diagnostic Test: Small RNA sequence — Comprehensive small RNA sequencing of serum or plasma-derived cf-tsRNAs to identify candidate biomarkers distinguishing HCC from NDC.
  Groups: HCC (Discovery, Small RNA-seq); Non-disease Control (Discovery, Small RNA-seq)
Diagnostic Test: Rt-qPCR — Construction of integrated cf- tsmiRNAs diagnostic classifier using machine learning
  Groups: HCC (Training, rt-qPCR); NDC (Training, rt-qPCR)
Diagnostic Test: Rt-qPCR — PCR-based validation of the tsRNA panel
  Groups: HCC (Testing, rt-qPCR); NDC (Testing, rt-qPCR)

SUMMARY:
Hepatocellular carcinoma (HCC) is often diagnosed at an advanced stage, and early detection is critical for improving patient outcomes. Despite this, reliable non-invasive biomarkers for early-stage HCC are limited.

This study seeks to develop a cell-free tsRNA (cf-tsRNA)-based liquid biopsy assay for accurate detection of early-stage HCC.

DETAILED DESCRIPTION:
Liver cancer is a major global health challenge, ranking as the 5th leading cause of cancer-related deaths in the U.S. and 3rd worldwide, with hepatocellular carcinoma (HCC) accounting for ~75% of cases. Incidence has more than tripled since 1980, and death rates have risen by ~2% annually, highlighting the need for improved detection and treatment. Prognosis remains poor: over 50% of HCC cases are diagnosed at stage IV, with a 1-year survival below 30%, whereas early-stage HCC (stages I-II) can achieve up to 74% 5-year survival with curative interventions. Major risk factors include viral hepatitis (HBV, HCV), alcohol abuse, obesity, type 2 diabetes, and non-alcoholic fatty liver disease (NAFLD), with non-viral HCC increasing in prevalence, particularly in Western countries. Screening programs target high-risk populations but miss many asymptomatic or average-risk individuals, contributing to late-stage diagnoses.

Biomarker discovery holds promise for improving early detection. Alpha-fetoprotein (AFP), the most widely used biomarker, has limited sensitivity for early-stage HCC (39-64%). tsRNAs (tRNA-derived small RNAs) are small, single-stranded RNA molecules derived from mature or precursor tRNAs that were first detected in the urine of patients with cancer in the 1970s. Emerging noninvasive markers offer complementary advantages: cell-free tsRNAs (cf-tsRNAs) are stable and highly sensitive for detection. Integrating these biomarker types could enable robust models for accurate early HCC detection, addressing a critical gap in clinical care.

This study seeks to validate a panel of more accurate and non-invasive biomarkers (cf-tsRNAs) in preoperative blood samples. Accurate early detection of HCC would help provide clear criteria for treatment decisions, such as timely surgical intervention or the addition of adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed diagnosis of hepatocellular carcinoma.
* Received standard diagnostic and staging procedures as per local guidelines
* Availability of at least one blood-derived sample, drawn before receiving any curative-intent treatment

Exclusion Criteria:

• Lack of or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who were diagnosed with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True Positive Rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True Negative Rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total number of cases (i.e.,accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Shao Y, Yu X, Zhou W, Yan J, Dong H, Ye G. Biological roles and potential clinical value of tRNA-derived small RNAs in gastrointestinal malignancies. Ann Med. 2025 Dec;57(1):2566866. doi: 10.1080/07853890.2025.2566866. Epub 2025 Oct 9. PMID 41069160
- [Background] Mao M, Chen W, Huang X, Ye D. Role of tRNA-derived small RNAs(tsRNAs) in the diagnosis and treatment of malignant tumours. Cell Commun Signal. 2023 Jul 21;21(1):178. doi: 10.1186/s12964-023-01199-w. PMID 37480078
- [Background] Lee S, Kim J, Valdmanis PN, Kim HK. Emerging roles of tRNA-derived small RNAs in cancer biology. Exp Mol Med. 2023 Jul;55(7):1293-1304. doi: 10.1038/s12276-023-01038-5. Epub 2023 Jul 10. PMID 37430089
- [Background] Zhou M, He X, Zhang J, Mei C, Zhong B, Ou C. tRNA-derived small RNAs in human cancers: roles, mechanisms, and clinical application. Mol Cancer. 2024 Apr 15;23(1):76. doi: 10.1186/s12943-024-01992-2. PMID 38622694
- [Background] Yuan J, Gu WC, Xu TX, Shen XJ, Li X, Shen L, Zhang Y, Ju SQ. 5'-transfer RNA halve-lysine-CTT as a promising biomarker for early detection of hepatocellular carcinoma. World J Gastrointest Oncol. 2025 Nov 15;17(11):111142. doi: 10.4251/wjgo.v17.i11.111142. PMID 41281472
- [Background] Sauzay C, Petit A, Bourgeois AM, Barbare JC, Chauffert B, Galmiche A, Houessinon A. Alpha-foetoprotein (AFP): A multi-purpose marker in hepatocellular carcinoma. Clin Chim Acta. 2016 Dec 1;463:39-44. doi: 10.1016/j.cca.2016.10.006. Epub 2016 Oct 11. PMID 27732875
- [Background] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Background] Xing H, Zheng YJ, Han J, Zhang H, Li ZL, Lau WY, Shen F, Yang T. Protein induced by vitamin K absence or antagonist-II versus alpha-fetoprotein in the diagnosis of hepatocellular carcinoma: A systematic review with meta-analysis. Hepatobiliary Pancreat Dis Int. 2018 Dec;17(6):487-495. doi: 10.1016/j.hbpd.2018.09.009. Epub 2018 Sep 15. PMID 30257796
- [Background] Choi JY, Jung SW, Kim HY, Kim M, Kim Y, Kim DG, Oh EJ. Diagnostic value of AFP-L3 and PIVKA-II in hepatocellular carcinoma according to total-AFP. World J Gastroenterol. 2013 Jan 21;19(3):339-46. doi: 10.3748/wjg.v19.i3.339. PMID 23372355
- [Background] Xu J, Chen B, Qi J, Wu J, Feng W, Jin K, Bao H, Chen L, Wang F. Evaluation of serum hsa_tsr014055 as a potential biomarker for diagnosis and prognosis of hepatocellular carcinoma. Ann Med. 2025 Dec;57(1):2528978. doi: 10.1080/07853890.2025.2528978. Epub 2025 Jul 6. PMID 40618217
- [Background] Jin K, Wu J, Yang J, Chen B, Xu J, Bao H, Zong W, Xie C, Chen L, Wang F. Identification of serum tsRNA-Thr-5-0015 and combined with AFP and PIVKA-II as novel biomarkers for hepatocellular carcinoma. Sci Rep. 2024 Nov 21;14(1):28834. doi: 10.1038/s41598-024-80592-y. PMID 39572775